CLINICAL TRIAL: NCT04804085
Title: Conduct of Anaesthesia During Acute Ischaemia Stroke: a Retrospective Case Series of Patients Undergoing Mechanical Thrombectomy
Brief Title: Anaesthesia for Mechanical Thrombectomy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 20AN004
Record Dates: First submitted 2020-11-09; First posted 2021-03-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Stroke, Ischemic; Anesthesia
Keywords: Anaesthesia; Ischaemic; Mechanical; Case Series; Endovascular; Thrombectomy; Stroke
MeSH Terms: conditions — Ischemic Stroke; Ischemia; Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Title: Conduct of anaesthesia during acute ischaemic stroke: a retrospective case series of patients undergoing mechanical thrombectomy.

Design: This study will be a retrospective consecutive observational case series

DETAILED DESCRIPTION:
The Aim of this study is to describe the baseline characteristics, procedural and post-operative clinical characteristics of anaesthetic care delivered to consecutive adult patients who underwent mechanical thrombectomy as part of their routine clinical care between 01/01/2016 and 01/10/2020 at Nottingham University Hospitals NHS Trust (sample size approximately 250).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Undergone mechanical thrombectomy for the management of acute ischaemia stroke between 01/01/2016-01/10/2020 at Nottingham University Hospitals NHS Trust.

Exclusion Criteria:

* No pre-specified exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be identified by existing clinical records of mechanical thrombectomy procedures undertaken at Nottingham University Hospitals and already collated as part of routine service evaluation and clinical care. Sampling will be consecutive. The sampling window (01/01/2016-01/10/2020) has been chosen because mechanical thrombectomy is a new therapy that was not undertaken in current form before 2016.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Evaluating the number of patients requiring mechanical thrombectomy | Through study completion, up to 9 months
  This retrospective study will identify the anaesthetic care delivered to a group of patients undergoing mechanical thrombectomy for the management of acute ischaemic stroke. The data collected will be from all patients that received this treatment between 01/01/2016 and 01/10/2020 at Nottingham University Hospitals NHS Trust. This data written up and of interest both to our organisation and to comparable neuroscience centres in the UK and internationally.
  Outcomes that will be measured in this clinical case study are highlighted below.

SECONDARY OUTCOMES:
Background information: Age (>/= 18 years of age) | Through study completion, up to 9 months
Background information: Gender (male or female) | Through study completion, up to 9 months
  Physiological gender
Background information: The degree of disability/dependence after a stroke will be measured using the presenting modified Rankin Score | Through study completion, up to 9 months
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.
Background information: Presenting blood pressure (systolic and diastolic) | Through study completion, up to 9 months
Background information: Presenting heart rate (beats per minute) | Through study completion, up to 9 months
Background information: The fitness of the patient will be measured using the American Society of Anaesthetists Classification | Through study completion, up to 9 months
  ASA I A normal healthy patient Healthy ASA II A patient with mild systemic disease ASA III A patient with severe systemic disease ASA IV A patient with severe systemic disease that is a constant threat to life ASA V A moribund patient who is not expected to survive without the operation ASA VI A declared brain-dead patient whose organs are being removed for donor purposes
Background information: Height of the patient (m) | Through study completion, up to 9 months
  BMI = Weight / (height x height)
Background information: Weight of the patient (kg) | Through study completion, up to 9 months
  BMI = Weight / (height x height)
Background information: Measuring the distance from referring hospital (miles) | Through study completion, up to 9 months
  Hospitals included: Kings Mill Hospital, Royal Derby Hospital, Leicester, Lincoln, Boston, Burton
The patient's stroke classification will be measured using National Institute for Health Stroke Scale | Through study completion, up to 9 months
  1-4 Minor stroke 5-15 Moderate stroke 16-20 Moderate to severe stroke 21-42 Severe stroke
Mode of anaesthesia | Through study completion, up to 9 months
  Awake / Sedated / Converted on-table to General Anaesthetic / GA.
To identify the anaesthetic agents used | Through study completion, up to 9 months
  Propofol / Alfentanil / Remifentanil / Fentanyl / Midazolam
The level of the anaesthetist (registrar / consultant) | Through study completion, up to 9 months
Intra - procedural observations: Measuring time spent with systolic blood pressure (mmHg) <10% of presenting BP (minutes) | Through study completion, up to 9 months
Intra - procedural observations: Quantifying any episodes of hypoxia (SpO2 <94%) | Through study completion, up to 9 months
Intra-procedural interventions: Identifying if the patient required vasopressors | Through study completion, up to 9 months
  None / metaraminol / ephedrine / noradrenaline
Measuring the response of treatment using the post-procedural Thrombolysis in Cerebral Infarction scale | Through study completion, up to 9 months
  Grade 0: no perfusion Grade 1: penetration with minimal perfusion Grade 2: partial perfusion Grade 2A: only partial filling (less than two-thirds) of the entire vascular territory is visualised Grade 2B: complete filling of all of the expected vascular territory is visualised but the filling is slower than normal Grade 3: complete perfusion
To identify the level of care required immediately post procedure (Level 0,1,2,3) | Through study completion, up to 9 months
Identify the duration of Intensive Care stays (days) | Through study completion, up to 9 months
Identify the duration of stay in hospital (days) | Through study completion, up to 9 months
  Whether in NUH or otherwise
To measure the long term outcome: National Institute for Health Stroke Scale at 24 hours post-procedure | Through study completion, up to 9 months
  1-4 Minor stroke 5-15 Moderate stroke 16-20 Moderate to severe stroke 21-42 Severe stroke
To measure the long term outcome: Modified Rankin Score at 90 days | Through study completion, up to 9 months
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.
To measure the long term outcome: Mortality at 90 days (survived / deceased) | Through study completion, up to 9 months
To measure the long term outcome: Discharge destination (home / institution) | Through study completion, up to 9 months

CONTACTS AND LOCATIONS:
Overall Officials: David Hewson (Consultant Anaesthetist), Principal Investigator — Nottingham University Hospitals Trust